CLINICAL TRIAL: NCT02658682
Title: Secondary Prevention of Depression Applying an Experimental Attentional Bias Modification Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: University of Oxford (Other); Sorlandet Hospital HF (Other Government); Diakonhjemmet Hospital (Other)
Responsible Party: Principal Investigator, Nils Inge Landrø, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NFR-229135
Record Dates: First submitted 2015-12-14; First posted 2016-01-20 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABM + (Experimental): Attention Bias Modification
  Interventions: Behavioral: Attention Bias Modification
- ABM - (Sham Comparator): Sham Attention Bias Modification
  Interventions: Behavioral: Sham Attention Bias Modification

INTERVENTIONS:
Behavioral: Attention Bias Modification — Computer based Attention Bias Modification
  Arms: ABM +
Behavioral: Sham Attention Bias Modification — Computer based Sham Attention Bias Modification
  Arms: ABM -

SUMMARY:
Depression (Major Depressive Disorder; MDD) has been dubbed "the common cold among the mental illnesses" and it is also a highly recurrent disorder. Secondary prevention has been identified as a key goal in the long-term management of depression. High recurrence rate suggests that there are specific vulnerability factors that increase people's risk for developing repeated episodes of the disorder. Preventive strategies should identify and ameliorate these factors to reduce the individual's risk of subsequent episodes. Biased attention for emotional stimuli is central to the cognitive model where increased sensitivity to negative cues is believed to fuel the negative thoughts and feelings in depression and play a key role in maintaining the illness. Selective biases in attention can be modified by a simple computerized technique; The Attention Bias Modification Task (ABM). This project aims to investigate whether ABM can reduce surrogate and clinical markers of relapse in a large group highly vulnerable to depressive episodes. The effects of ABM, immediately after the two weeks intervention, on three key risk factors for depression will be studied: Residual symptoms, cortisol awakening response and emotion regulation strategies. The participants will be followed up after 1 month, 6 months and 12 months. The hypothesis that ABM will reduce subsequent episodes of low mood over the following 12 months in this group in a manner predicted by early changes in these risk factors will be investigated. It will also be tested if such effects in the lab may be dependent on candidate genes which affect serotonin reuptake and which have been implicated in malleability and emotional learning. Effects on underlying neural correlates of emotion regulation will be studied in an fMRI experiment in a sub-sample and which will also be stratified by serotonin transporter genotype (see also NCT02931487). The predictive value of meta cognitions related to rumination and the possible mediating effects of automatic thoughts and perceived stress will also be investigated in a sub group (see also NCT02648165).

The characterization of the cognitive, genetic and neural mechanisms underlying the ABM effect will have key implications for future treatment development and combination with other treatment modalities like pharmacotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Nondepressed subjects (based on the MINI structured interview) with a history of major depression

Exclusion Criteria:

* Current or past neurological illness, bipolar disorder, psychosis or drug addiction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in residual symptoms of depression. Self report. | At baseline and immediately after ABM intervention (during first week after ABM).
  Beck Depression Inventory
Change in residual symptoms of depression. Clinician rating | At baseline and immediately after ABM intervention (during first week after ABM).
  Hamilton Depression Rating Scale

SECONDARY OUTCOMES:
Recurrence of major depressive episodes | Will be measured 12 month after baseline
  Measured by the MINI structured interview
Changes in Emotion Regulation | At baseline.
  Emotion Regulation Questionnaire (ERQ).
Changes in Rumination | At baseline and 12 months after intervention
  The Rumination Response Scale
Changes in cortisol response. | At baseline, immediately after ABM intervention and one month after intervention.
  Cortisol samples from saliva measured by diural variation (6 samples).
Changes in symptoms of anxiety | At baseline, immediately after ABM intervention (during first week after ABM intervention), 1 month after intervention, 6 months after intervention and 12 months after intervention
  Beck Anxiety Inventory

OTHER OUTCOMES:
Automatic thoughts | At baseline, immediately after ABM intervention (average one day), 1 month after intervention, 6 months after intervention and 12 months after intervention
  Automatic Thought Questionnaire (ATQ)
Changes in perceived stress | At baseline, immediately after ABM intervention (average one day), , 1 month after intervention, 6 months after intervention and 12 months after intervention
  Perceived Stress Scale (PSS).
Meta cognitions | At baseline and 12 months after intervention
  Positive and Negative Beliefs about Rumination scale (PBRS and NBRS)
5-HTTLPR+A>G polymorphic variation divided by the triallelic functional "high expressive" versus "low expressive" genotype will moderat the effect of ABM on residual symptoms compared to neutral ABM placebo condition | Immediately after ABM intervention.
Brain Derived Neurotrophic Factor (BDNF) val66met polymorphic variation linked to Brian Derived Neurotrophic Factor (BDNF) variation will moderate the effect of ABM on residual symptoms compared to neutral ABM placebo condition | Immediately after ABM intervention.
A serotonergic cumulative Genetic score, including (5-HHTLPR, HTR1A 8rs6295) and HTR 2A (rs 6311) polymorphisms will moderate the effects of ABM on residual symptoms compared to neutral placebo condition | Immediately after ABM intervention.
Change in residual symptoms of depression. Self report | One month after intervention, 6 months after intervention and 12 months after intervention
  Beck Depression Inventory
Change in residual symptoms of depression. Clinical rating | One month after intervention, 6 month after intervention and 12 month after intervention
  Hamilton Depression Rating Scale
Primary outcome measures will be modified by the degree of attentional change during the ABM intervention. | Immediately after the ABM intervention
Primary outcome measures will be modified by executive functioning | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nils I Landrø, Dr. Phil, Principal Investigator — University of Oslo
Locations (2):
- Norway (2):
  - Sørlandet Hospital, Department of Psychiatry, Arendal, Aust-Agder
  - University of Oslo, Department of Psychology, Oslo

REFERENCES:
- [Derived] Bo R, Kraft B, Skilbrei A, Jonassen R, Harmer CJ, Landro NI. Inhibition moderates the effect of attentional bias modification for reducing residual depressive symptoms: A randomized sham-controlled clinical trial. J Behav Ther Exp Psychiatry. 2024 Dec;85:101982. doi: 10.1016/j.jbtep.2024.101982. Epub 2024 Aug 2. PMID 39111231
- [Derived] Bo R, Kraft B, Jonassen R, Pedersen ML, Harmer CJ, Landro NI. The long-term effects of ABM on symptom severity in patients with recurrent depression: A randomized sham-controlled trial. J Affect Disord. 2023 Nov 1;340:886-892. doi: 10.1016/j.jad.2023.08.024. Epub 2023 Aug 12. PMID 37579884
- [Derived] Bo R, Kraft B, Jonassen R, Harmer CJ, Hilland E, Stiles TC, Haaland VO, Aspesletten MEB, Sletvold H, Landro NI. Symptom severity moderates the outcome of attention bias modification for depression: An exploratory study. J Psychiatr Res. 2021 Jun;138:528-534. doi: 10.1016/j.jpsychires.2021.04.027. Epub 2021 May 5. PMID 33984807
- [Derived] Jonassen R, Harmer CJ, Hilland E, Maglanoc LA, Kraft B, Browning M, Stiles TC, Haaland VO, Berge T, Landro NI. Effects of Attentional Bias Modification on residual symptoms in depression: a randomized controlled trial. BMC Psychiatry. 2019 May 8;19(1):141. doi: 10.1186/s12888-019-2105-8. PMID 31068158